CLINICAL TRIAL: NCT00003862
Title: A Phase II Trial of Preoperative Chemotherapy and Chemoradiotherapy for Potentially Resectable Adenocarcinoma of the Stomach
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9904; CDR0000067026
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2003-09

CONDITIONS: Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Fluorouracil; Leucovorin; Paclitaxel; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: leucovorin calcium
Drug: paclitaxel
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy and radiation therapy in treating patients who have stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of preoperative chemoradiotherapy in patients with potentially resectable adenocarcinoma of the stomach.
* Determine the pathologic response rate, curative resection rate, and survival in patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.

OUTLINE: Patients receive fluorouracil IV over 24 hours on days 1-21, cisplatin IV over 1 hour on days 1-5, and leucovorin calcium IV over 15 minutes on days 1, 8, 15, and 22. A second course is administered beginning on day 29.

Chemoradiotherapy begins at the end of the second course of chemotherapy and 1 week of rest (day 57). Patients receive fluorouracil IV over 24 hours 5 days a week concurrently with radiotherapy for 5 weeks and paclitaxel IV over 3 hours once weekly during these 5 weeks on days 1, 8, 15, 22, and 29.

Approximately 4-5 weeks after chemoradiotherapy, patients with no evidence of metastatic disease undergo surgical resection.

Patients are followed every 3 months for 1 year, every 6 months for 5 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 21-49 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the stomach

  * Stage IB, II, IIIA, IIIB, and IV (T2-3, any N, M0)

    * No lymph node metastases outside the field of resection (e.g., supraclavicular, mediastinal, or paraaortic nodes)
  * Potentially resectable
  * May involve the gastroesophageal junction, but bulk of tumor must be in the stomach
  * No distant metastases
  * No pleural or pericardial effusion
* No peritoneal disease diagnosed by laparoscopy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 16 weeks

Hematopoietic:

* Absolute granulocyte count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No hypertension

Neurologic:

* No cerebrovascular disease
* No diabetic neuropathy
* No mental status abnormalities

Other:

* No uncontrolled diabetes
* No infection
* No other malignancies within past 5 years except resected squamous cell or basal cell skin cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to stomach

Surgery:

* No prior surgery to stomach

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A. Ajani, MD, Study Chair — M.D. Anderson Cancer Center
Locations (55):
- United States (55):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Medical Center, Concord, California
  - Northridge Hospital Medical Center, Northridge, California
  - University of California Davis Cancer Center, Sacramento, California
  - Penrose - St. Francis Health Services, Colorado Springs, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Lutheran General Hospital Cancer Care Center, Park Ridge, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - Porter Memorial Hospital, Valparaiso, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - McLaren Regional Cancer Center, Flint, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Inc., Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Harrington Cancer Center, Amarillo, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Result] Ajani JA, Winter K, Okawara GS, Donohue JH, Pisters PW, Crane CH, Greskovich JF, Anne PR, Bradley JD, Willett C, Rich TA. Phase II trial of preoperative chemoradiation in patients with localized gastric adenocarcinoma (RTOG 9904): quality of combined modality therapy and pathologic response. J Clin Oncol. 2006 Aug 20;24(24):3953-8. doi: 10.1200/JCO.2006.06.4840. PMID 16921048
- [Result] Okawara GS, Winter K, Donohue JH, et al.: A phase II trial of preoperative chemotherapy and chemoradiotherapy for potentially resectable adenocarcinoma of the stomach (RTOG 99-04). [Abstract] J Clin Oncol 23 (Suppl 16): A-4019, 312s, 2005.